CLINICAL TRIAL: NCT04060784
Title: Maxillary Anterior Immediate Tooth Replacement With and Without Socket-shield: a One Year Prospective Study
Brief Title: Maxillary Anterior Immediate Tooth Replacement With and Without Socket-shield
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: Nobel Biocare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5190036
Record Dates: First submitted 2019-08-16; First posted 2019-08-19 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Anterior Teeth
Keywords: Immediate implant placement and provisionalization; Socket shield technique; Root shield; Soft tissue level change; Soft tissue volume change; IIPP; SST
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Intervention Model Description: There are two groups in this study, 13 patients each. Subjects who fulfill the inclusion criteria with one failing anterior tooth will be included into this study.
Who Masked: Outcomes Assessor
Masking Description: Data analysis will be blind. Intraexaminer reliability will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Immediate implant placement and provisionalization (Experimental): On the control group, Implant will be placed immediately after tooth extraction. The gap between the implant and buccal bone will be filled with bone graft. Temporary crown will be attached to implant fixture.
  Interventions: Procedure: Immediate implant placement and provisionalization
- Socket shield technique (Experimental): On the test group, Implant will be placed immediately after tooth extraction. A piece of root shield will be retained intentionally at facial side. Temporary crown will attached to implant fixture.
  Interventions: Procedure: Immediate implant placement and provisionalization

INTERVENTIONS:
Procedure: Immediate implant placement and provisionalization — Failing tooth will be extracted and immediate placed endosseous implant
  Other Names: Socket shield technique

SUMMARY:
The purpose of this clinical controlled study is to compare anterior facial gingival level change between Immediate implant placement and provisionalization with bone graft and with socket shield technique.

DETAILED DESCRIPTION:
Immediate implant placement and provisionalization, short for IIPP, is one of a very viable option for failing anterior teeth. It has been advocated with documented success for more than 20 years. Despite the decent results, the challenges remains on the altered of the facial implant tissue architecture. To avoid the facial contour change and the possible following esthetic problem, clinicians have tried several ways to preserve the contour, like bone grafting in the gap between the facial bone and implant, or enhance facial gingival tissue thickness through augmentation procedures.

The concept of retaining part of the root, or root shield in conjunction with IIPP was proposed around 8 to 9 years ago. So-called socket shield technique. It has claimed to have successfully preserve the facial contour. Animal studies and couple clinical studies have showed decent results.

The purpose of this clinical controlled study is to compare the facial gingival level change between IIPP with bone graft and with socket shield technique. There are two groups in this study, 13 patients each. Extrusion criteria including male under 21 years old, female under 23 years old, smoker, pregnant patient, history of head and neck radiation, soft tissue defect like inflammation, recession, active infection. On the control group, patient will received IIPP with bone graft; On the test group, IIPP and socket shield technique will be provided. All clinical examinations and data collections will be performed by one investorgator, who will do the measurement at presurgical appointment, Tps, the time of implant placement, Tm0, 6-months Tm6, and 12-months after implant placement Tm12. Data analysis will be blind. Intraexaminer reliability will be performed.

We are looking at 12 elements in this study. The main variable will be facial gingival level change. We will use Intraoral scanner and the 3D images obtained at different time point will be superimposed, to see if there is any significant change between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 21 years of age or older and able to consent to treatment.
* Good oral hygiene. Patient's oral hygiene should be control to a certain level before start the procedure: Plaque Index (PI) score19 ≤20% and Papillary Bleeding Index (PBI) score20 of less than 5%
* Have a single failing maxillary anterior tooth with periodontally healthy adjacent teeth.
* No active infection associated with the failing tooth
* An extraction socket that will allow a facial implant-socket space of ≥2mm after placement of an implant with a minimum dimensions of 3.0 mm diameter and 13.0 mm in length.
* Presence of opposing dentition (natural teeth, fixed or removable prostheses)

Exclusion Criteria (control group)

* Systemic disease and/or associated medications that could interfere with implant therapy.
* Dental history of bruxism, parafunction habit, and/or lack of stable posterior occlusion.
* Smoker.
* History of head and neck radiation.
* Pregnant patient, intending to conceive or breast feeding.
* Soft tissue defect (inflammation, tissue cleft, recession, papilla loss, unhealthy tissue) around a future implant site.

Exclusion Criteria (test group)

* Systemic disease and/or associated medications that could interfere with implant therapy.
* Dental history of bruxism, parafunction habit, and/or lack of stable posterior occlusion.
* Smoker.
* History of head and neck radiation.
* Pregnant patient, intending to conceive or breast feeding.
* Soft tissue defect (inflammation, tissue cleft, recession, papilla loss, unhealthy tissue) around a future implant site.
* Teeth with active infection like periodontal disease, periapical lesions.
* Teeth with vertical root fractures on the buccal aspect, horizontal fracture at or below buccal bone level.
* Teeth with any other pathologies affecting the buccal part of the root, like external or internal resorptions.
* History of head and neck radiation.
* Any mobility of the extraction tooth.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Facial gingival level change | At baseline (pre-op) and at 12 months after surgery
  The baseline measurement will be compared with digital superimposition of intraoral scanned images at 12 months post-op

SECONDARY OUTCOMES:
Soft tissue volume change | At baseline (pre-op) and 12 months after surgery
  The baseline measurement will be compared with digital superimposition of intraoral scanned images at 12 months post-op

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Kan, DDS, Principal Investigator — Loma Linda dental implant department
Locations (2):
- United States (2):
  - Loma Linda University school of dentistry, Loma Linda, California
  - Loma Linda University Health, Loma Linda, California

IPD SHARING:
Plan to Share IPD: Undecided